CLINICAL TRIAL: NCT03198273
Title: The Efficacy of Clinical Pilates Exercises on Individuals With Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülşan Taşpınar, physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EasternMediterranianUniversity
Record Dates: First submitted 2017-06-02; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Lumbar Disc Herniation
Keywords: clinical pilates; exercise; lumbar disc herniation; chronic low back pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pilates exercises (Experimental): Participants will exercise 3 times a week for 6 weeks (18 sessions in total, 45-60 minutes each session) in accompany with a physiotherapist. Since the chosen model for exercise training is clinical pilates exercises, separate patient training will be needed. First 3 weeks planned as Warming Phase, Exercise Phase (first 3 weeks), Cooling Phase; and Second 3 weeks planned as Warming Phase, Exercise Phase (first 3 weeks), Cooling Phase.
  Interventions: Other: Clinical pilates exercises
- Physiotherapy Program (Experimental): Standard physiotherapy program consisting of conservative treatment is applied to both groups. The conservative treatment schedule to be applied to planned as 10 sessions, 3 times a week.
  Interventions: Other: physiotherapy program

INTERVENTIONS:
Other: Clinical pilates exercises — servical, lumbal, pelvic muscles
  Other Names: exercise program
  Arms: Clinical pilates exercises
Other: physiotherapy program — hot-pack will apply for 20 minutes. Convansionel TENS will apply on the lumbar regions of the cases of the control group paravertebrally with
  Other Names: standart physiotherapy program
  Arms: Physiotherapy Program

SUMMARY:
The aim of the study is to determine the effects of clinical Pilates Exercises on the level of pain, functional status, flexibility, static and dynamic endurance of the truncus muscles and quality of life in patients with lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, between the ages of 30-60,
* Have been diagnosed according to Magnetic Resonance Imaging results, in one or several of the levels of L3-L4 / L4-L5 / L5-S1 in the case of Bulging and Protuberance lumbar disc hernia,
* At least 6 weeks with back and leg pain,
* Those who will be able to participate in the exercise program regularly,
* Those who are not included in the physiotherapy program in the last 6 months,,
* With mental, auditory and visual problems that will prevent communication will be included in the study.

Exclusion Criteria:

* Individuals, with spinal stenosis,
* Having previously described lumbar spine surgery,
* Having severe neurological deficits,
* Having primary or metastatic spinal malignancy,
* Having vascular problem at a later stage in the lower extremity,
* Diagnosed with osteoporosis,
* Those who are pregnant,
* Having uncontrolled hypertension,
* With anger-dependent anguish will not be included in the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | nine weeks
  Visual Analogue Scale (VAS) is a pain intensity measurement scale with validity and reliability. The patient will be told that they can evaluate their pain from 0 to 10 on a 10 cm horizontal line. It will be explained that if there is no pain, 0 (the leftmost point), the most severe pain will be 10 (the rightmost point). According to these explanations, patients will be asked to mark their pain intensity on a 10 cm chart. On the 10 cm chart, the distance between the point marked by the patient and the leftmost 0 will be measured by the ruler and the value will be recorded.

SECONDARY OUTCOMES:
Functional Level Status | nine weeks
  The Oswestry Lumbar Scale (ODI) was developed by Fairbank to assess functional impairment. There are 10 questions evaluating various daily activities of this scale and 6 options for each question between 0-5. In this scale, the degree of clinical pain severity, personal care, lifting, walking, sitting, standing, sleeping, social life, travel and change degree of the pain are questioned. The minimum score taken from the scale is 0, the maximum score is 50. 0-4 points mean there is no disability, 5-14 points are mild, 15-24 points are moderate, 25-30 points are severe and 35-50 points are considered to be complete functional disability.
Quality of Life Level | nine weeks
  Short Form-36 (SF-36) will assess the health-related quality of life of individuals. The form consists of a total of 36 articles which can be filed by the patient. The scale consists of 8 subscales related to health. Physical function (10 articles), social function (2 articles), role limitations due to physical problems (3 articles), role limitations due to emotional problems (3 articles), mental health (5 articles), fitness (4 articles), pain (2 articles), general health [general overview point (5 articles) and health change (1 article)]. The scores from each subscale range from 0-100. 0 indicates the worst condition and 100 the best health condition. The SF-36 is suitable for personal evaluation, and can be applied to people over 14 years of age or face to face computerized or trained personnel.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyrenia 7/24 Orthopedics and Traumatology Clinic, Kyrenia, Karakum, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taspinar G, Angin E, Oksuz S. The effects of Pilates on pain, functionality, quality of life, flexibility and endurance in lumbar disc herniation. J Comp Eff Res. 2023 Jan;12(1):e220144. doi: 10.2217/cer-2022-0144. Epub 2022 Dec 1. PMID 36453667